CLINICAL TRIAL: NCT06335329
Title: Point-of-Care Ultrasound Findings and Impact on Vaping Behaviors in Adolescents
Brief Title: Point-of-Care Ultrasound (POCUS) Findings and Impact on Vaping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00133616
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Vaping
Keywords: vaping; Point-of-care ultrasound; adolescents; POCUS
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants will be randomized on a 1:1 ratio to be able to see and discuss their ultrasound results, or remain blinded to them.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard vaping cessation counseling (SOC) + ultrasound (US) (Active Comparator): Participants will receive SOC via a publicly available infographic from the Food and Drug Administration). They will also be provided with a discussion of lung US findings
  Interventions: Behavioral: Discussion of point-of-care ultrasound lung findings
- Standard vaping cessation counseling (SOC) alone (No Intervention): Participants will receive a SOC alone. They will be kept blinded to their lung point-of-care ultrasound findings and will not be able to visualize the images as the ultrasound is performed.

INTERVENTIONS:
Behavioral: Discussion of point-of-care ultrasound lung findings — The investigator will obtain point-of-care ultrasound images to assess the lung findings in 12 lung fields. These 12 lung fields will include the standard protocol of the upper and lower halves of the anterior, lateral, and posterior chest bilaterally. Subjects' ultrasound images will be scored using a modified lung ultrasound score (LUS). Each of the 12 lung fields will be scored from 0-5, with a total score of 0-60 (noted below). The participants will watch their ultrasound being performed, looking at their lungs in real time. Then, the ultrasound findings will be discussed with the participant.
  Modified LUS 0: No B-lines present
  1. 1 well-defined B-line
  2. 2-3 well-defined B-lines
  3. >3 B-lines
  4. Confluent B-lines
  5. Lobar consolidation
     * C: Noted if subpleural consolidation present
     * E: Noted if pleural effusion present
  Arms: standard vaping cessation counseling (SOC) + ultrasound (US)

SUMMARY:
Vaping has emerged as a prominent public health crisis in recent years. In 2023, the National Youth Tobacco Survey found that more than 2.1 million adolescents endorse vaping, with 25% of those endorsing daily use. Many adolescents also perceive vapes as safer than cigarettes, and more acceptable to use both indoors and outdoors compared to cigarettes. Vapes are available in numerous device and delivery systems, with the psychoactive agent commonly including nicotine or cannabis, although these can be of a wide variety of concentrations and formulations. They may be ultra-compact and allow for ease of concealment. In addition, they are produced in a variety of appealing flavorings such as candy, desserts, and fruits. Other constituents include the liquids and aerosolized components of the vaping cartridges, including formaldehyde, acetone, glycerol, propylene glycol, acetaldehyde, and heavy metals. Many of the flavoring concentrates, as well as the vaporized solvents, have not been evaluated for long term safety. One of these additives, vitamin E acetate, present in primarily illicit vaping devices, rose to national attention in 2019 for a suspected link to the dramatic increase in vaping/e-cigarette associated lung injury (EVALI) cases, with over 60 confirmed deaths since that time.

To our knowledge, there are no studies evaluating the lung ultrasound findings of asymptomatic vapers. However, there is data to suggest that vaping can lead to pulmonary toxicity in in-vitro and animal models, including increased inflammatory cytokines, hyperreactivity, and oxidative stress. In addition, studies found the risk of bronchitic symptoms is twice as likely in current adolescent vapers, compared to those who have never vaped before. Given the potential pulmonary toxicity of vaping, as well as the increased percentage of adolescent vaping activity in recent years, investigators aim to evaluate baseline lung ultrasound findings in adolescents who vape. Concurrently, investigators will assess if observing their lung ultrasound findings can alter their attitudes and behaviors towards vaping. Prior adult studies have found that showing patients' their atherosclerosis plaque increased the motivation to quit and cessation rates. Additionally, data in pregnant patients found real-time ultrasound feedback of smoking effects on the fetus lead to near abstinence in light smokers. Given the frequent use of point-of-care ultrasound in the emergency department, investigators hope to assess an innovative intervention for cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-18 years of age
* Has own individual cell phone or email for communication
* Member of a vaping history group that is not yet full for enrollment (ex: up to 100 vapers, up to 100 non-vapers)
* Able to speak and understand English

Exclusion Criteria:

* Chronic Lung Disease
* History of pneumothorax
* Prior thoracic surgery including VATS (Video-assisted thoracoscopic surgery)
* Sickle cell disease
* Current or prior cancer
* Significant congenital heart disease
* Acute upper respiratory infection (cough or congestion in the last 3 days)
* Acute chest trauma
* Acute pulmonary embolism
* Sedation medication administered prior to study image acquisition
* Known allergy or sensitivity to ultrasound gel
* Significant acute psychosis, mania, or suicidal ideation
* Any other medical or psychiatric condition or other significant concern that in the investigator's opinion would impact participant safety or compliance with study instructions, or potentially confound the interpretation of findings
* Inability or unwillingness of subject or legal guardian/representative to give informed consent/assent.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Lung Ultrasound Findings | Day 1
  The purpose of this study is to establish the lung findings in vaping adolescents, specifically point-of-care ultrasound scores, and to identify factors such as age, sex, race, and vital signs, that contribute to variability in lung findings. Each of the 12 lung fields will be scored from 0-5, with a total score of 0-60. The modified LUS is defined below.
  Modified LUS 0: No B-lines present
  1. 1 well-defined B-line
  2. 2-3 well-defined B-lines
  3. >3 B-lines
  4. Confluent B-lines
  5. Lobar consolidation
     * C: Noted if subpleural consolidation present
     * E: Noted if pleural effusion present
Behavioral Changes | Day 1, at 2 weeks, at 2 months
  Questionnaire to assess if observing lung findings can alter adolescents' vaping behaviors, risk perception, behavioral intent, and motivation to quit.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Gorukanti A, Delucchi K, Ling P, Fisher-Travis R, Halpern-Felsher B. Adolescents' attitudes towards e-cigarette ingredients, safety, addictive properties, social norms, and regulation. Prev Med. 2017 Jan;94:65-71. doi: 10.1016/j.ypmed.2016.10.019. Epub 2016 Oct 20. PMID 27773711
- [Background] Overbeek DL, Kass AP, Chiel LE, Boyer EW, Casey AMH. A review of toxic effects of electronic cigarettes/vaping in adolescents and young adults. Crit Rev Toxicol. 2020 Jul;50(6):531-538. doi: 10.1080/10408444.2020.1794443. Epub 2020 Jul 27. PMID 32715837
- [Background] Fadus MC, Smith TT, Squeglia LM. The rise of e-cigarettes, pod mod devices, and JUUL among youth: Factors influencing use, health implications, and downstream effects. Drug Alcohol Depend. 2019 Aug 1;201:85-93. doi: 10.1016/j.drugalcdep.2019.04.011. Epub 2019 May 23. PMID 31200279